CLINICAL TRIAL: NCT00045318
Title: A Phase I Study of DX-8951f (Exatecan Mesylate for Injection) in Patients With Renal Dysfunction
Brief Title: Exatecan Mesylate in Treating Patients With Advanced Solid Tumors and Kidney Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DAIICHI-8951A-PRT026; UCLA-0201008; CDR0000256866 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2103
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2003-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of exatecan mesylate in treating patients who have advanced solid tumors and kidney dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of exatecan mesylate in patients with advanced solid tumors and varying degrees of renal dysfunction.
* Determine the dose-limiting and non-dose-limiting toxic effects of this drug in these patients.
* Determine the effects of renal dysfunction on the plasma pharmacokinetics and pharmacodynamics of this drug in these patients.
* Establish a model for dosing this drug in patients with impaired renal function.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to severity of renal dysfunction (normal vs mild vs moderate vs severe).

Patients receive exatecan mesylate IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients in each renal dysfunction stratum receive escalating doses of exatecan mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients in the normal renal function stratum do not undergo dose escalation.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 45 patients (6 normal, 9 mild, 12 moderate, and 18 severe renal dysfunction) will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor refractory to standard therapy or for which no standard therapy exists
* Renal function as defined by the following parameters:

  * Normal (creatinine clearance (CrCl) greater than 80 mL/min)
  * Mild dysfunction (CrCl 50-80 mL/min)
  * Moderate dysfunction (CrCl 30-50 mL/min)
  * Severe dysfunction (CrCl less than 30 mL/min)
  * End-stage renal disease (requiring dialysis)
* No symptomatic or active brain metastases (e.g., edema or progression on CT scan or MRI)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin normal
* AST or ALT no greater than 2 times upper limit of normal
* Albumin at least 2.8 g/dL

Renal

* See Disease Characteristics

Cardiovascular

* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction within the past 6 months

Other

* No concurrent serious infection
* No other life-threatening illness
* No overt psychosis or mental disability or other incompetency that would preclude informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea) and recovered
* No prior exatecan mesylate
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy
* Concurrent megestrol for appetite stimulation allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery

* At least 4 weeks since prior major surgery and recovered
* No concurrent anticancer surgery

Other

* At least 4 weeks since prior investigational drugs including analgesics or antiemetics
* At least 1 week since prior grapefruit juice
* No other concurrent anticancer therapy
* No other investigational drugs during and for 4 weeks after study
* No concurrent grapefruit juice
* No other concurrent anticancer cytotoxic therapy
* Concurrent chronic hemodialysis or ambulatory peritoneal dialysis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - St. Luke's Lutheran Hospital, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas